CLINICAL TRIAL: NCT02970981
Title: A Pilot Trial of Ipilimumab With Nivolumab for Participants With Resected Stages IIIB/IIIC/ IV Melanoma
Brief Title: Study of Combination of Ipilimumab and Nivolumab in Patients With Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-00098
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Melanoma
Keywords: Monoclonal antibody; Programmed Death-1 (PD-1); Programmed Death-Ligand 1 (PD-L1); Cytotoxic T lymphocyte-associated antigen 4 (CTLA-4); Antigen
MeSH Terms: conditions — Melanoma; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab and Ipilimumab (Experimental): Dosing during cycle 1 will consist of: 3 mg/kg of Nivolumab+ Ipilimumab at 1 mg/kg. Each induction treatment cycle is comprised of 4 doses of Nivolumab and 4 doses of Ipilimumab given every three weeks for a total of 12 weeks (cycle 1)
  Dosing during cycles 2-5 will consist of flat dose Nivolumab at 480 mg every 4 weeks (Q4W) for 48 weeks.
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab
  Other Names: Opdivo; NSC 748726
Biological: Ipilimumab
  Other Names: Yervoy; NSC 732442

SUMMARY:
The purpose of this study is to assess the safety and tolerability of treatment with Nivolumab in combination with Ipilimumab in subjects with resected Stages IIIB/IIIC/ IV melanoma.

DETAILED DESCRIPTION:
The investigators hypothesize that PD-1 blockade combined with CTLA-4 blockade using ipilimumab would have a favorable effect on the expansion and activity of human CD8+ T cytotoxic lymphocytes (CTLs) specific for tumor-associated antigens (ie, self antigens), which would translate into improved anti-cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 16 years of age;
* Histologic diagnosis of resected Stages IIIB/IIIC/ IV melanoma, with no evidence of disease clinically and radiologically, and negative surgical margins. All melanomas regardless of primary site of disease will be allowed;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Prior chemotherapy or immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer) must have been completed at least 4 weeks before study drug administration, and all adverse events have either returned to baseline or stabilized;
* Prior treated brain or meningeal metastases must be without magnetic resonance imaging (MRI) evidence of progression for at least 8 weeks and off immunosuppressive doses of systemic steroids (> 10 mg/day prednisone or equivalent) for at least 2 weeks before study drug administration;
* Prior systemic radiation therapy must have been completed at least 4 weeks before study drug administration. Prior focal radiotherapy completed at least 2 weeks before study drug administration. No radiopharmaceuticals (strontium, samarium) within 8 weeks before study drug administration;
* Immunosuppressive doses of systemic medications, such as steroids or absorbed topical steroids (doses > 10 mg/day prednisone or equivalent) must be discontinued at least 2 weeks before study drug administration;
* Completed nitrosourea treatment at least 6 weeks before administration of any study drug;
* Prior surgery that required general anesthesia must be completed at least 4 weeks before study drug administration. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before study drug administration and subjects should be recovered;
* Screening laboratory values must meet the following criteria:

white blood cells (WBCs) ≥ 2000 cells/μL

* neutrophils ≥ 1500 cells/μL
* platelets ≥ 100 x 103/μL
* hemoglobin ≥ 9.0 g/dL
* serum creatinine ≤ 2 mg/dL
* AST ≤ 2.5 x upper limit of normal (ULN) without, and ≤ 5 x ULN with hepatic metastasis
* ALT ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis
* bilirubin ≤ 2 x ULN (except subjects with Gilbert's syndrome, who must have total bilirubin < 3.0 mg/dL)
* Females of childbearing potential must:
* use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab.
* For female subjects to be considered as not having childbearing potential, they must meet 1 or more of the following criteria:
* postmenopausal for at least 24 consecutive months;
* surgically sterile (ie, have had a hysterectomy or bilateral oophorectomy);
* females with irregular menstrual periods and/or on hormone replacement therapy must have a documented serum follicle stimulating hormone level > 35 mIU/mL;
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception.
* Subject must have read, understood, and provided written informed consent and HIPAA authorization after the nature of the study has been fully explained; and
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Subjects who fulfill any of the following conditions at Screening will not be eligible for admission into the study:
* History of severe hypersensitivity reactions to other mAbs;
* Prior non-melanoma malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix or breast;
* Subjects with any active autoimmune disease (Appendix 3) or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy;
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS);
* Positive tests for hepatitis B virus surface antigen (HBV SAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection;
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PDL-2, or anti-CTLA-4 antibody (or any other antibody targeting T cell co-stimulation pathways);
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids;
* Underlying medical condition (eg, a condition associated with diarrhea) that, in the Investigator's opinion, would make the administration of either study drug or both study drugs hazardous to the subject or obscure the interpretation of toxicity determination or adverse events;
* Pregnant or nursing; or
* Current participation in another clinical study involving treatment with medications, radiation or surgery, or prior participation in this study.
* Patients are excluded if they have active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for [lowest minimum is 4 weeks or more] after treatment is complete and within 28 days prior to the first dose of nivolumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.

As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen.

* Allergies and Adverse Drug Reaction

  1. History of allergy to study drug components
  2. History of severe hypersensitivity reaction to any monoclonal antibody

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2022-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Weber, MD, PhD, Principal Investigator — NYU Perlmutter Cancer Center
Locations (1):
- Laura and Isaac Perlmutter Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Khushalani NI, Vassallo M, Goldberg JD, Eroglu Z, Kim Y, Cao B, Ferguson R, Monson KR, Kirchhoff T, Amato CM, Burke P, Strange A, Monk E, Gibney GT, Kudchadkar R, Markowitz J, Brohl AS, Pavlick A, Richards A, Woods DM, Weber J. Phase II clinical and immune correlate study of adjuvant nivolumab plus ipilimumab for high-risk resected melanoma. J Immunother Cancer. 2022 Nov;10(11):e005684. doi: 10.1136/jitc-2022-005684. PMID 36450385

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 participants were enrolled in the study; 2 participants were deemed ineligible before starting the study.
Groups:
- Nivolumab and Ipilimumab: Dosing during cycle 1 will consist of: 3 mg/kg of Nivolumab+ Ipilimumab at 1 mg/kg. Each induction treatment cycle is comprised of 4 doses of Nivolumab and 4 doses of Ipilimumab given every three weeks for a total of 12 weeks (cycle 1)
  Dosing during cycles 2-5 will consist of flat dose Nivolumab at 480 mg every 4 weeks (Q4W) for 48 weeks.
  Nivolumab
  Ipilimumab
Period: Overall Study
Arm/Group | Nivolumab and Ipilimumab
Started | 16
Received Intervention | 16
Completed Induction Therapy (4 Cycles) | 15
Completed Maintenance Therapy (48 Weeks) | 14
Completed | 14
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab and Ipilimumab
Number analyzed (Participants) | 16
Age, Customized [Count of Participants; unit: Participants]
  >= 16 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Disease Stage at Entry [Count of Participants; unit: Participants] — CT scans with contrast of the chest, abdomen, and pelvis as well as MRI scans of the brain with gadolinium were done for disease evaluation. The earliest stage melanomas are stage 0 (melanoma in situ), and then range from stages I (1) through IV (4). As a rule, the lower the number, the less the cancer has spread. A higher number, such as stage IV, means cancer has spread more. And within a stage, an earlier letter means a lower stage.
  Participants
    IIIB | 6
    IIIC | 5
    IV | 4
    IIB | 1

OUTCOME MEASURES:

1. Primary Outcome: Relapse-Free Survival
Description: Number of participants who are relapse-free at 48 months after initiating treatment in the study.
Time Frame: Month 48 Post-Treatment Initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and Ipilimumab
Number analyzed (Participants) | 16
Participants | 12

2. Secondary Outcome: Number of Cases of Adverse Events Occurring During Study
Description: The adverse events are evaluated per Common Terminology Criteria for Adverse Events (CTCAE) V4.
Time Frame: Month 12 Post-Treatment Initiation
Measure: Number; unit: cases of adverse events
Arm/Group | Nivolumab and Ipilimumab
Number analyzed (Participants) | 16
cases of adverse events | 238

3. Secondary Outcome: Overall Survival
Description: Percentage of participants who are alive at at 48 months after initiating treatment in the study.
Time Frame: Month 48 Post-Treatment Initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and Ipilimumab
Number analyzed (Participants) | 16
Participants | 16

ADVERSE EVENTS:
Time Frame: 48 weeks post-treatment
Arm/Group | Nivolumab and Ipilimumab
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 5/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab and Ipilimumab (N=16)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab and Ipilimumab (N=16)
Abdominal Pain (Gastrointestinal disorders) | 3
Increase in alanine aminotransferase (Hepatobiliary disorders) | 3
Increase in Alkalina Phosphatase (General disorders) | 1
Allergic rhinitis (General disorders) | 2
Anemia (Blood and lymphatic system disorders) | 4
Anorexia (Psychiatric disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Blurred vision (General disorders) | 2
Chest wall discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Chills (General disorders) | 3
Conjunctivitis (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Increase in Creatinine (Metabolism and nutrition disorders) | 1
Dehydration (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
Dry mouth (General disorders) | 2
Green floater in eye (Eye disorders) | 1
Edema (Blood and lymphatic system disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 2
Fever (General disorders) | 2
GERD (Gastrointestinal disorders) | 2
Loose stool (Gastrointestinal disorders) | 7
Alopecia (General disorders) | 1
Malaise (General disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Cramping (Musculoskeletal and connective tissue disorders) | 2
Hernia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Nasal congestion (General disorders) | 5
Non productive cough (General disorders) | 1
Nausea (General disorders) | 6
General pain (General disorders) | 9
Papulopostular rash (Skin and subcutaneous tissue disorders) | 3
Decrease in platelet count (Blood and lymphatic system disorders) | 1
Productive cough (General disorders) | 2
Pruritis (Skin and subcutaneous tissue disorders) | 16 (17)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 16 (30)
Sore throat (Infections and infestations) | 3
Urinary urgency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT02970981/Prot_SAP_000.pdf